CLINICAL TRIAL: NCT05508438
Title: A Prospective, Multicenter, Objective Performance Criteria Clinical Study to Evaluate the Efficacy and Safety of the Transfemoral Mitral Valve Repair System in the Treatment of Patients With Moderately Severe and Severe Functional Mitral Regurgitation(FMR)
Brief Title: To Evaluate the Efficacy and Safety of the Transfemoral Mitral Valve Repair System in the Treatment of Patients With Moderately Severe and Severe Functional Mitral Regurgitation(FMR) Who Remained Clinically Symptomatic After Guideline-directed Medical Treatment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pan Xiangbin (Other)
Responsible Party: Sponsor-Investigator, Pan Xiangbin, Chief, Department of Structural Heart DiseaseAffiliation, Chinese Academy of Medical Sciences, Fuwai Hospital
Organization: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KOKA-2021-02
Record Dates: First submitted 2022-07-21; First posted 2022-08-19 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Mitral Valve Insufficiency
Keywords: Heart Valve Disease; Cardiovascular Diseases
MeSH Terms: conditions — Mitral Valve Insufficiency; Heart Valve Diseases; Cardiovascular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Other)
  Interventions: Device: Transfemoral mitral-valve repair

INTERVENTIONS:
Device: Transfemoral mitral-valve repair — Transfemoral mitral-valve repair

SUMMARY:
To confirm the effectiveness and safety of the transcatheter mitral valve repair system for the treatment of chronic moderate to severe (3+) or severe (4+) functional mitral regurgitation (FMR) who remained clinically symptomatic after guideline-directed medical treatment.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, objective performance criteria clinical design.Patients are moderate to severe (3+) or severe (4+) functional mitral regurgitation (FMR) who remained clinically symptomatic after guideline-directed medical treatment. All subjects receive clinical follow-up immediately after procedure, before discharge, 30 days after procedure, 6 months after transfemoral mitral-valve repair, 12 months and 2 yeas，3 years，4 years after Transfemoral mitral-valve repair.

The primary outcome is defined as all-cause death and rehospitalization due to heart failure 12 months after Transfemoral mitral-valve repair.

The secondary outcomes include：Rate of rehospitalization due to heart failure after operation；Rate of postoperative mitral regurgitation (MR ≤ 2+)；Rate of New York Heart Association (NYHA) Function Class I or II after Transfemoral mitral-valve repair；Change in 6 minutes walk test distance；Improvement value of quality of life changes assessed by Kansas City Cardiomyopathy Questionnaire (KCCQ)；Echocardiographic changes in left ventricular end diastolic volume (LVEDV) from baseline；Acute procedural success，Acute device success.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age ≥ 18 yrs；
* 2. Symptomatic functional mitral regurgitation (FMR) (≥3+) due to ischemic or non-ischemic cardiomyopathy

Note 1: Functional MR requires the presence of overall or localized left ventricular wall motion abnormalities that are considered to be the primary cause of MR. Despite the eligibility, subjects may not enroll if leaflet prolapse or other evidence of degenerative MR is present.

Note 2: An Eligible transthoracic echocardiography must be obtained at least 30 days after the subject has been stabilized on optimal therapy with Guideline Directed Medical Therapy (GDMT), or at least 30 days under the following conditions after meeting two of the following conditions：Coronary revascularization and/or implantation of a cardiac resynchronization therapy device (CRT-P or CRT-D) or reprogramming of the implanted CRT-P or CRT-D resulting in an increase in biventricular pacing (from <92% to ≥92%).

* 3. Subjects have been adequately treated according to applicable criteria, including treatment for coronary artery disease, left ventricular dysfunction, mitral regurgitation, and heart failure (e.g., with cardiac resynchronization therapy (CRT or CRT-D), coronary revascularization, and/or have received stable GDMT, confirmed by the local heart team;
* 4. NYHA functional class II to IV;
* 5. Left ventricular ejection fraction (LVEF) ≥20%;
* 6. Left ventricular end-systolic dimension (LVESD) ≤ 70 mm;
* 7. The subject's mitral valve is anatomically suitable for mitral valve repair;
* 8. Elevated BNP >150 pg/ml or corrected NT-proBNP ≥600 pg/ml or heart failure hospitalization within the past 12 months ('corrected' refers to a 4% reduction in the BNP or NT-proBNP cutoff for every increase of 1 kg/m2 in BMI above a reference BMI of 20 kg/m2);
* 9. After evaluation, the femoral vein approach is suitable and the puncture through atrial septum is feasible;
* 10. The subjects have been informed of the nature of this study, understand the purpose of the clinical trial, and voluntarily participate in and sign the informed consent form.

Exclusion Criteria:

* 1) Echocardiographic evidence of intracardiac mass, thrombus, or vegetation;
* 2) The presence of other severe heart valve disease requiring surgical intervention.;
* 3) After mitral valve surgery or mitral valve transcatheter surgery;
* 4)Hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis, infiltrative cardiomyopathy (e.g., amyloidosis, hemochromatosis, sarcoidosis, etc.), or any other structural heart disease causing heart failure other than dilated cardiomyopathy of either ischemic or non-ischemic etiology.;
* 5) Autoimmune myocarditis;
* 6) Heart failure caused by tachyarrhythmia is effective after GDMT treatment;
* 7) Moderate to severe right heart dysfunction or an estimated pulmonary artery systolic pressure (PASP) > 70 mmHg assessed by echocardiography;
* 8) History of acute myocardial infarction in the prior 4 weeks or untreated clinically significant coronary artery disease requiring revascularization;
* 9) Any percutaneous cardiac intervention within the 30 days, or any cardiac surgery within the 6 months prior to randomization, or any implant of any Cardiac Resynchronization Therapy (CRT-P) or Cardiac Resynchronization Therapy with cardioverter-defibrillator (CRT-D) or Implantable Cardioverter Defibrillator (ICD) within the last 30days prior to subject registration，or patients who meet the indications of CRT-P and CRT-D but are not implanted;
* 10) In the judgment of the investigator, the subject's femoral vein is unable to accommodate a 22F catheter or has an ipsilateral deep venous thrombosis; or the anatomy is not accessible for transseptal puncture;
* 11)) Subjects in whom transesophageal echocardiography (TEE) or general anesthesia is contraindicated;
* 12) End-stage heart failure (ACC/AHA stage D), or prior orthotopic heart transplantation, or on the waiting list for heart transplantation.；
* 13) Active endocarditis; Or valvular degeneration caused by active rheumatic heart disease or rheumatic disease (such as poor compliance, perforation, etc)；
* 14) Severe Chronic Obstructive Pulmonary Disease (COPD) (requiring continuous home oxygen therapy or long-term application of steroid hormone medication)；
* 15) Cerebrovascular accident within 30 days prior to randomization or symptomatic severe carotid stenosis (> 70% by ultrasound), carotid artery stenting within 30 days.；Cerebrovascular accident (hemorrhagic) within 6 months；
* 16) History of acute peptic ulcer or gastrointestinal bleeding within 3 months；
* 17)Hemorrhagic or coagulopathic disorders, contraindications to antithrombotic medication；
* 18) Modified Rankin Scale ≥4.；
* 19) The subjects suffer from diseases that may lead to difficulty in evaluating treatment (e.g., cancer, severe metabolic disease, psychosis, etc.)；
* 20）Pregnant or breastfeeding women, or women who plan to become pregnant within the next 12 months.

Note: Women of childbearing age should take a pregnancy test with a negative result within 14 days prior to registration and use scientifically safe contraception；

* 21) Hemodynamic instability defined as systolic pressure < 90 mmHg without afterload reduction, cardiogenic shock, or the need for inotropic support or an intra-aortic balloon pump；
* 22) Active infections requiring antibiotic therapy (in the case of temporary illness, antibiotics must be discontinued for at least 14 days before the subject can be enrolled).；
* 23) Currently participating in an investigational drug or another device study that has not completed its primary endpoints or would clinically interfere with the endpoint of this study. Note: Trials requiring extended follow-up for products that were investigational, but have since become commercially available, are not considered investigational trials；
* 24) In the judgment of the investigator, subjects may not complete the trial according to poor compliance or in other circumstances when the investigator determines that the subject is unfit to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-08-30 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
The composite endpoint of all-cause mortality and rehospitalization due to heart failure 12 months after Transfemoral mitral-valve repair | 12 months after Transfemoral mitral-valve repair
  All-cause mortality and rehospitalization due to heart failure

SECONDARY OUTCOMES:
rehospitalization | 30 days,6 months,12months after Transfemoral mitral-valve repair
  The rate of rehospitalization due to heart failure
postoperative | 30 days,6 months,12months after Transfemoral mitral-valve repair
  The rate of postoperative mitral regurgitation (MR ≤ 2+)
New York Heart Association (NYHA) | 30 days,6 months,12months after Transfemoral mitral-valve repair
  The rate of New York Heart Association (NYHA) Function Class I or II.
walk test | 12 months after Transfemoral mitral-valve repair
  Change in 6-minutes walk test distance.
Kansas City Cardiomyopathy Questionnaire (KCCQ) | 12 months after Transfemoral mitral-valve repair
  Improvement value of quality of life changes assessed by Kansas City Cardiomyopathy Questionnaire (KCCQ)
left ventricular end diastolic volume (LVEDV) | 12 months after Transfemoral mitral-valve repair
  Echocardiographic changes in left ventricular end diastolic volume (LVEDV) from
procedural success | Before discharge
  Acute procedural success
device success | Immediately after procedure
  Acute device success

CONTACTS AND LOCATIONS:
Overall Officials: Xiangbin Pan, MD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Structral Heart Disease Center, Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li H, Chen Y, Zhang J, Guo Y, Guo Q, Guo H, Gong J, Ni D, Wang F, Xue W, Duan F. TEERAI-Pre: A Multiview Artificial Intelligence Model for Preoperative Assessment of Transcatheter Edge-to-Edge Mitral Valve Repair Using Multiview, Multimodal Echocardiography. J Am Heart Assoc. 2026 Jan 30:e044333. doi: 10.1161/JAHA.125.044333. Online ahead of print. PMID 41614293